CLINICAL TRIAL: NCT04162626
Title: New Families- Innovation and Development of the Child Health Services in Oslo
Acronym: NF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VID Specialized University (Other)
Collaborators: Oslo Municipality (Other Government); University of Oslo (Other); Norwegian Institute of Public Health (Other Government); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kari Glavin, Professor, VID Specialized University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/1378
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Primary Prevention
Keywords: public health nurse; intervention; home visit
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Supportive home visits by public health nurses to new parents from 28 weeks in pregnancy until the child is two years.
  Interventions: Other: Supportive home visits to new families
- Control (Other): Follow up as usual at the Child health center
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Supportive home visits to new families — The new families are offered home visits by a public health nurse from 28 weeks in pregnancy until the child is two years old. The number of home visits depends on the families needs and wishes. They also get the usual follow up from the Child health center.
  Arms: Intervention
Other: Treatment as usual — Follow up at the Child health center according to national regulations
  Arms: Control

SUMMARY:
The New Families (NF) program will improve quality of existing services, secure personalised service and early intervention in Child Health Service (CHS) in Oslo. The study will measure the effects of a primary prevention family-centered healthcare intervention in Norwegian CHS.

DETAILED DESCRIPTION:
The New Families (NF) program will improve quality of existing services, secure personalised service and early intervention in Child Health Service (CHS) in Oslo. The study will: 1) Measure the effects of a primary prevention family-centered healthcare intervention in Norwegian CHS, 2) Create case studies from CHS praxis advancing Public Health Nurse (PHN) training and education in Oslo and Norway, 3) Establish a model for how to include users in service development in CHS, 4) Enhance the knowledge base of the PHN practice in CHS Anticipated results: The project will bolster the knowledge base for education and professional practices within the service by strengthen the existing research within the field. The anticipated results of the project are that the intervention will increase maternal and parental self-efficacy, reduce the risk of postpartum depression among first-time mothers, reduce parental stress, increase social support, improve maternal attachment, improve generic health status, improve partner relationship and improve child development compared with usual care. The intervention research in this project can be a future model for service improvement in the CHS.

ELIGIBILITY:
Inclusion Criteria:

* First time parents living in the chosen districts

Exclusion Criteria:

* All other parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Depression in mothers in pregnancy | 28 weeks pregnancy
  Edinburgh postnatal depression scale (EPDS). 10 items. Score 0-30. Score 12 or above indicate postpartum depression.
Depression in fathers when partner is pregnant | 28 weeks pregnancy
  Edinburgh postnatal depression scale (EPDS). 10 items. Score 0-30. Score 12 or above indicate postpartum depression.
Depression in mothers three months postpartum | 3 months postpartum
  Edinburgh postnatal depression scale (EPDS). 10 items. Score 0-30. Score 12 or above indicate postpartum depression.
Depression in fathers three months postpartum | 3 months postpartum
  Edinburgh postnatal depression scale (EPDS). 10 items. Score 0-30. Score 12 or above indicate postpartum depression.
Sense of Coherence in mothers in pregnancy | 28 weeks pregnancy
  Sense of Coherence Scale (SOC 13). 26 items. Score 13-90. Higher score is positive, score under 66 is low.
Sense of Coherence in fathers in pregnancy | 28 weeks pregnancy
  Sense of Coherence Scale (SOC 13). 26 items. Score 13-90. Higher score is positive, score under 66 is low.
Sense of Coherence in mothers three months postpartum | 3 months postpartum
  Sense of Coherence Scale (SOC 13). 26 items. Score 13-90. Higher score is positive, score under 66 is low.
Sense of Coherence in fathers three months postpartum | 3 months postpartum
  Sense of Coherence Scale (SOC 13). 26 items. Score 13-90. Higher score is positive, score under 66 is low.
Self-Efficacy in mothers 6 weeks postpartum | 6 weeks postpartum
  Perceived Maternal Parenting Self-Efficacy (PMP S-E) 20 items. score 22-88. A higher score indicates a higher level of maternal self-efficacy
Self-Efficacy in fathers 6 weeks postpartum | 6 weeks postpartum
  Perceived Maternal Parenting Self-Efficacy (PMP S-E) 20 items. score 22-88. A higher score indicates a higher level of maternal self-efficacy
Self-Efficacy in mothers 3 months postpartum | 3 months postpartum
  Perceived Maternal Parenting Self-Efficacy (PMP S-E) 20 items. score 22-88. A higher score indicates a higher level of maternal self-efficacy
Self-Efficacy in fathers 3 months postpartum | 3 months postpartum
  Perceived Maternal Parenting Self-Efficacy (PMP S-E) 20 items. score 22-88. A higher score indicates a higher level of maternal self-efficacy
Parental Stress in fathers 3 months postpartum | 3 months postpartum
  Parental Stress Scale (PSS) is formatted in the form of an 18-item self-report scale. Items represent positive (e.g. emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood. A higher score indicates a higher level of parental stress.
Parental Stress in mothers 3 months postpartum | 3 months postpartum
  Parental Stress Scale (PSS) is formatted in the form of an 18-item self-report scale. Items represent positive (e.g. emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood. A higher score indicates a higher level of parental stress.
Quality of Life in women and men during pregnancy and postpartum | Pregnancy week 28, 3 months postpartum, 12 months postpartum.
  To explore first-time parents' QoL during pregnancy and first-time mothers QoL postpartum, and to evaluate the difference in QoL between mothers in the intervention and control districts. Instrument: WHOQOL-BREF, 26-item. Score 4-20, higher scores indicate higher QoL.

SECONDARY OUTCOMES:
What are the barriers and facilitators to implementation of the PHN intervention? | The interviews will take place about 12 months postpartum
  This research question will be explored by addressing the process of implementation.
  Data will be collected through a short survey and semi-structured interviews with PHNs and users (first-time mothers/fathers).
  An interview guide will be developed

CONTACTS AND LOCATIONS:
Overall Officials: Kari Glavin, PhD, Principal Investigator — VID Specialized University
Locations (1):
- VID Specialized University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There will be four doctoral students (PhD) in the project

REFERENCES:
- [Derived] Brekke M, Smastuen MC, Glavin K, Amro A, Solberg B, Oygarden AU, Saether KM, Haugland T. The impact of New Families home visiting program on first-time mothers' quality of life and its association with social support: a non-randomized controlled study. BMC Public Health. 2023 Dec 8;23(1):2457. doi: 10.1186/s12889-023-17285-0. PMID 38066502

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04162626/Prot_SAP_000.pdf